CLINICAL TRIAL: NCT04139564
Title: Safety and Effectiveness of Virtual Reality Utilizing EaseVRx for the Reduction of Chronic Pain and Opioid Use
Brief Title: EaseVRx for the Reduction of Chronic Pain and Opioid Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AppliedVR Inc. (Industry)
Collaborators: Geisinger Clinic (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-1017; 5R44DA050231 (NIH)
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EaseVRx group (Experimental): Each subject will be asked to complete a 56-day program using the EaseVRx virtual reality headset with assigned modules each week. Each week, subjects will be asked to complete 7 modules (one per day), each approximately 5 minutes in duration, for a total of 56 modules across the program.
  Interventions: Device: EaseVRx headset
- Active control group VR Sham (Active Comparator): Each subject will be asked to complete a program accessible via VR that includes 2d visual wildlife scenes similar to some EaseVRx content
  Interventions: Device: Active control VR sham program

INTERVENTIONS:
Device: EaseVRx headset — EaseVRx is a virtual reality therapy intended to treat chronic pain
  Arms: EaseVRx group
Device: Active control VR sham program — VR, 2d visual wildlife scenes similar to some EaseVRx content
  Arms: Active control group VR Sham

SUMMARY:
EaseVRx, a software-based virtual reality (VR) medical device, is intended to offer users a prescription pain management tool that manages the symptoms associated with chronic pain and reduces or eliminates the risk of opioid dependence. The investigators will conduct a proof-of-concept randomized study to assess the feasibility and efficacy of using EaseVRx as a 56-day, VR-based, at-home program among 100 chronic low back pain patients by gathering pilot data on the efficacy of the intervention in decreasing pain, reducing opioid/non-opioid pharmacotherapy, and improving pain-related quality of life.

DETAILED DESCRIPTION:
EaseVRx, a software-based virtual reality (VR) medical device, is intended to offer users a prescription pain management tool that manages the symptoms associated with chronic pain and reduces or eliminates the risk of opioid dependence. EaseVRx is based on principles of cognitive behavioral therapy, pain psychology, mindfulness-based stress reduction, biofeedback, and distraction therapy commonly used in interdisciplinary pain rehabilitation programs. The investigators will conduct a proof-of-concept randomized study to assess the feasibility and efficacy of using EaseVRx as a 56-day, VR-based, at-home program among 100 chronic low back pain patients by gathering pilot data on the efficacy of the intervention in decreasing pain, reducing opioid/non-opioid pharmacotherapy, and improving pain-related quality of life. While VR has been tested in academic medical centers and shown to be efficacious in the management of acute pain, this study will investigate the feasibility of VR use at home to manage chronic pain in preparation for a larger efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Low back pain experienced ≥ 3 days per week on average for ≥ 6 months
* Pre-medication NPRS score ≥ 5 stable for ≥ 3 months

Exclusion Criteria:

* Exclusions based on potential medical or lifestyle confounders:

  * Has a body mass index (BMI) > 40 kg/m2
  * Pain related to cancer, fibromyalgia, or disk herniation
  * History of a major psychiatric disorder not controlled with medication or has behavioral factors that would interfere with proper study procedures
  * Is not ambulatory/has significant motor impairment
  * Surgery in the past 3 months
  * Open workers compensation claim
  * Planning to have surgery in the next 3 months
  * Planning to start a new exercise program in the next 3 months
  * Planning to start a new treatment for their pain (e.g. medication, physiotherapy, acupuncture, electrical nerve stimulation) in the next 3 months
* Exclusions based on potential drug-related cofounders:

  * Current or recent history (in past year) of substance abuse disorder
  * Currently pregnant/breastfeeding or planning to in the next 3 months
  * Was administered an epidural steroid during the 3 months prior to screening
* Exclusions based on ability to use EaseVR effectively:

  * Comorbidities including neurological, psychosocial, sensory, or other disorders that may impact pain perception
  * Diagnosis of epilepsy, dementia, migraines, or other neurological disorders that may prevent VR usage, and/or other medical conditions predisposed to nausea and dizziness
  * Hypersensitivity to flashing lights or motion
  * Claustrophobia
  * Lack of stereoscopic vision
  * Severe hearing impairment
  * Injury to eyes, face, or neck that prevents comfortable VR usage
  * Planning to take a vacation from their home for more than one week in the next 8 weeks

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chulhyun Ahn, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Medical Center, Danville, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EaseVRx Group | Active Control Group VR Sham
Started | 52 | 55
Completed | 52 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EaseVRx Group | Active Control Group VR Sham | Total
Number analyzed (Participants) | 52 | 55 | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 55 | 107
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (13.5) | 51.4 (12.9) | 51.4 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 40 | 78
  Male | 14 | 15 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 50 | 52 | 102
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Numerical Pain Rating Scale [Mean (Standard Deviation); unit: units on a scale from 0 to 10] — The scale ranges from 0 to 10 with larger numbers implying greater pain.
  units on a scale from 0 to 10 | 6.0 (1.9) | 5.9 (1.5) | 5.9 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Pain: Numerical Pain Rating Scale
Description: Numerical Pain Rating Scale; scale from 0 to 10 with higher numbers implying greater pain
  The outcome values presented below are the difference between baseline pain and pain at 12 weeks. Specifically, baseline pain score minus 12 week pain score
  A positive difference implies that pain was reduced
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EaseVRx Group | Active Control Group VR Sham
Number analyzed (Participants) | 52 | 55
units on a scale | 0.6 (1.67) | 1.3 (1.49)

2. Secondary Outcome: Number of Outcome Assessments Completed by Participant
Description: Thirty four assessments were attempted. This measure notes the total number of assessments completed by each participant
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: total number of assessments completed
Arm/Group | EaseVRx Group | Active Control Group VR Sham
Number analyzed (Participants) | 51 | 53
total number of assessments completed | 30 (14.3) | 28 (15.7)

3. Secondary Outcome: Patient Compliance
Description: number of VR modules completed. For the EaseVRx group this would be the number of EaseVRx modules completed with worst 0 - 56 best. For the Active control VR Sham group this would be the number of ShamVR modules completed with worst 0 - 56 best.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: modules
Arm/Group | EaseVRx Group | Active Control Group VR Sham
Number analyzed (Participants) | 50 | 48
modules | 37 (18.4) | 40 (19.3)

4. Secondary Outcome: Opioid Consumption
Description: Morphine Milligram Equivalents (MME)
Time Frame: 12 weeks
Measure: Geometric Mean (Standard Error); unit: Morphine Milligram Equivalents(MME)
Arm/Group | EaseVRx Group | Active Control Group VR Sham
Number analyzed (Participants) | 45 | 50
Morphine Milligram Equivalents(MME) | 6.75 (3.37) | 5.67 (2.56)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | EaseVRx Group | Active Control Group VR Sham
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/55
Other Adverse Events (participants affected / at risk) | 0/52 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/64/NCT04139564/Prot_SAP_000.pdf